CLINICAL TRIAL: NCT00503035
Title: Molecular Targeting of 15-LOX-1 for Apoptosis Induction in Human Colorectal Cancers
Brief Title: Molecular Targeting of 15-Lipoxygenase-1 (15-LOX-1) for Apoptosis Induction in Human Colorectal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM02-592; NCI-2012-01522 (Registry Identifier: NCI CTRP); 1R01CA106577-01A1 (NIH); NCT00258219 (obsolete NCT alias)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial Adenomatous Polyposis; Colorectal Tumors; Molecular Targeting; Celecoxib; Celebrex; SC-58635; Apoptosis Induction; Colon; Rectum; colonoscopy; Biopsy
MeSH Terms: conditions — Adenomatous Polyposis Coli; Colorectal Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Celecoxib (Experimental): Celecoxib 400 mg orally twice daily for 6 months. Up to 23 additional colon tissue biopsies (the size of a pencil tip), additional 20 minutes on colonoscopy procedure.
  Interventions: Drug: Celecoxib; Procedure: Colonoscopy Biopsy

INTERVENTIONS:
Drug: Celecoxib — 400 mg by mouth twice daily x 6 months
  Other Names: Celebrex; SC-58635
Procedure: Colonoscopy Biopsy — Up to 23 additional colon tissue biopsies (the size of a pencil tip), additional 20 minutes on colonoscopy procedure

SUMMARY:
Primary Objective:

* To determine whether celecoxib downregulates GATA-6 expression to upregulate 15-LOX-1 expression and induce apoptosis in human rectal tumors, researchers will measure GATA-6 and 15-LOX-1 expression, 13-S-HODE levels, and apoptosis rates in normal and colorectal polyp epithelial tissues before and after 6 months of celecoxib treatment of patients with familial adenomatous polyposis (FAP).

DETAILED DESCRIPTION:
Celecoxib is a drug that was developed to treat arthritis. However, celecoxib may also help to stop or slow the growth of colon and rectal tumor cells.

At the start of the study, you will be asked questions about your medical history, have a complete physical exam, and have around 2 tablespoons of blood drawn for blood tests as part of your routine care for familial adenomatous polyposis. Also, blood tests such as fasting blood glucose and lipid profiling (cholesterol, LDL, HDL and triglyceride) will be assessed to determine eligibility. Women who are able to have children must have a negative blood pregnancy test within 14 days of starting celecoxib.

Before your scheduled colonoscopy, you will fill out a form asking about any medications and nutritional supplements that you are taking. In addition, you will be asked to complete a diet history. This will help researchers to evaluate patients' dietary habits. The questionnaire takes about 15 minutes to complete. You will also have around 1 teaspoon of blood drawn to measure the amount of celecoxib in your blood. Then, during your already scheduled colonoscopy procedure, you will have additional tissue biopsies (the size of a pencil tip) of your colon taken. For a colonoscopy procedure, a flexible tube with a light attached to the end is used to look inside your colon/lower gut. The biopsies will be taken through the flexible tube using a special cutting tool. Up to 23 biopsy samples may be taken. The biopsies should take about 20 extra minutes to complete.

After the procedure, you will start taking celecoxib by mouth once every 12 hours for 6 months. You will also have around 1 teaspoon of blood drawn to measure the amount of celecoxib in your blood at the completion of month 2 and 4 of celecoxib treatment. At the end of the 6 month treatment period, you will have another colonoscopy procedure. This is an additional procedure performed solely for this study and is not part of your standard of care for the treatment of familial adenomatous polyposis. A second set of biopsies will be taken (23 maximum). These biopsy samples will be studied and compared to the samples taken before treatment with celecoxib. You will also have around 1 teaspoon of blood drawn to measure the amount of celecoxib in your blood.

You will be contacted by phone 72 hours after your first dose of celecoxib and then every 2 weeks for the study to check for any side effects you may be experiencing.

The maximum amount of time you will remain on this study is 6 months. If at any time, you experience any intolerable side effects, you will be taken off the study.

This is an investigational study. Celecoxib is FDA approved and commercially available for familial adenomatous polyposis patients to reduce polyp formation. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of familial adenomatous polyposis (patients should have colorectal remnant that can be biopsied. Patients who have had total colorectal surgical resection are not eligible).
2. Adequate bone marrow function (ANC > 1500 ml, platelet count > 100,000/ml). Serum creatinine, total bilirubin, and ALT < 1.5 upper limit normal.
3. Over 16 years of age.
4. Patient is able to give an informed consent.
5. Women of childbearing potential (women are considered to be of childbearing potential unless they are at 2 or more years post-menopausal/or surgically sterile), must:

   * Not be pregnant or lactating.
   * use adequate contraceptive measures (abstinence, IUD, birth control pills, or diaphragm or condom with spermicidal gel) starting with last menses and throughout the study duration.
   * Have a negative serum pregnancy test within 14 days of starting celecoxib.

Exclusion Criteria:

1. Inflammatory bowel disease.
2. Intake of anti-inflammatory medications (e.g., non-steroidal, aspirin, and sulfasalazine) that cannot be discontinued starting 3 days prior to the enrollment.
3. Chemotherapy or radiation therapy in less than three months from the time of enrollment.
4. Individuals who are taking Coumadin that can not be discontinued starting 7 days prior to the enrollment.
5. Individuals who have received an investigational chemopreventive agent during the month prior to the biopsies.
6. History of bleeding diathesis.
7. History of sulfonamides (sulfa) allergies.
8. History of cardiovascular diseases that might include the following: myocardial infarction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery.
9. Uncontrolled hypertension (> 135/> 85 mm Hg on three repeated measurements during the 6 weeks prior to enrollment on the study).
10. Diagnosis of diabetes.
11. Smoking history during the 6 months prior to enrollment on the study.
12. Uncontrolled hypercholesteremia (low-density lipoprotein cholesterol (LDL-C) > 130). Hypercholesteremia needs to be controlled following the updated the National Cholesterol Education Program Adult Treatment Panel III Guidelines for at least 3 months prior to enrollment on the study. Hypercholesteremia treatment needs to be continued during the enrollment on the protocol.
13. Family history of premature coronary disease (i.e., onset < 55 years of age).
14. Metabolic syndrome diagnosis in patients who are 30 years or older. (The diagnosis of metabolic syndrome is made when three or more of these risk factors are present):

    * Waist circumference: Men > 102 cm (> 40 in); Women > 88 cm (> 35 in). *Triglycerides = 150 mg/dl (= 1.69 mmol/L).
    * High-density lipoprotein cholesterol (HDL-C): [Men < 40 mg/dl (< 1.03 mmol/L), Women <50 mg/dl (< 1.29 mmol/L)].
    * Blood pressure = 130/= 85 mm Hg.
    * Fasting glucose = 110 mg/dl (= 6.1 mmol/L).
15. History of deep venous thrombosis, pulmonary embolism, systemic lupus erythematous, family history of protein S or C deficiencies or prior heparin-induced thrombocytopenia.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-08-20 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Shureiqi, MD, Principal Investigator — M.D. Anderson Cancer Center; Robert S. Bresalier, MD, Study Chair — M.D. Anderson Cancer Center; Patrick Lynch, MD, JD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Lynch PM, Morris JS, Ross WA, Rodriguez-Bigas MA, Posadas J, Khalaf R, Weber DM, Sepeda VO, Levin B, Shureiqi I. Global quantitative assessment of the colorectal polyp burden in familial adenomatous polyposis by using a web-based tool. Gastrointest Endosc. 2013 Mar;77(3):455-63. doi: 10.1016/j.gie.2012.11.038. Epub 2013 Jan 18. PMID 23332604
- [Background] Yang P, Zuo X, Advani S, Wei B, Malek J, Day RS, Shureiqi I. Celecoxib Colorectal Bioavailability and Chemopreventive Response in Patients with Familial Adenomatous Polyposis. Cancer Prev Res (Phila). 2022 Apr 1;15(4):217-223. doi: 10.1158/1940-6207.CAPR-21-0066. PMID 34610992
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 participants consented, 4 participants were inevaluable.
Groups:
- Celecoxib: Celecoxib 400 mg orally twice daily for 6 months. Up to 23 colon tissue biopsies (the size of a pencil tip).
Period: Overall Study
Arm/Group | Celecoxib
Started | 47
Completed | 27
Not Completed | 20
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 3
Not completed — Ineligible | 15

BASELINE CHARACTERISTICS:
Population: 29 patients completed 6 months of celecoxib treatment
Arm/Group | Celecoxib
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: 13-HODE Colonic Tissue Levels
Description: 13-HODE colonic tissue levels measured by Liquid chromatography and tandem mass spectrometry measurements (LC/MS/MS) in colorectal normal and polyp tissues
Time Frame: Baseline to post 6 months of celecoxib treatment
Measure: Mean (Standard Deviation); unit: ng/mg tissue protein
Groups:
- Celecoxib: Celecoxib 400 mg orally twice daily for 6 months. Up to23 additional colon tissue biopsies (the size of a penciltip), additional 20 minutes on colonoscopy procedure.
  Celecoxib: 400 mg by mouth twice daily x 6 months Colonoscopy Biopsy: Up to 23 additional colon tissuebiopsies (the size of a pencil tip), additional 20 minuteson colonoscopy procedure
Arm/Group | Celecoxib
Number analyzed (Participants) | 27
ng/mg tissue protein
  polyps before celecoxib treatment | 14.56 (9.93)
  polyps after celecoxib treatment | 18.83 (14)
  Normal: before celecoxib treatment | 23.02 (18.55)
  Normal: after celecoxib treatment | 20.03 (11.7)

2. Secondary Outcome: PGE2 Colonic Tissue Levels
Description: PGE2 colonic tissue levels measured by Liquid chromatography and tandem mass spectrometry measurements (LC/MS/MS) in colorectal normal and polyp tissues
Time Frame: at the baseline colonoscopy (or sigmoidoscopy in patients who had undergone colectomy) before the initiation of celecoxib, and the follow-up colonoscopy or sigmoidoscopy was performed after celecoxib treatment (month 6)
Measure: Mean (Standard Deviation); unit: ng/mg tissue protein
Groups:
- Celecoxib: Celecoxib 400 mg orally twice daily for 6 months. Up to 23 additional colon tissue biopsies
Arm/Group | Celecoxib
Number analyzed (Participants) | 27
ng/mg tissue protein
  Polyps: before celecoxib treatment | 14.71 (6.95)
  Polyps: after celecoxib treatment | 20.62 (10.48)
  Normal: before celecoxib treatment | 21.48 (14.32)
  Normal: after celecoxib treatment | 24.99 (18.25)

ADVERSE EVENTS:
Time Frame: Study subjects were contacted by phone 72 hr. after the first celecoxib doses and every 2 weeks thereafter for the rest of the celecoxib treatment duration for toxicity assessment. In addition, subjects had evaluation for toxicity as part of history and physical during a clinical visit at the end of the treatment, at 6 months
Description: Adverse events accessed for the participants who received celecoxib for any duration on the study.
Arm/Group | Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=32)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=32)
Abdominal pain (Gastrointestinal disorders) | 5
Allergic Reaction (Skin and subcutaneous tissue disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 4
Blurred vision (Eye disorders) | 1
Bruising (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Cramping (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Flatulance (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Oral Ulceration (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 2
Rectal hematoma (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hot flashes (General disorders) | 2
Increase appetite (Gastrointestinal disorders) | 2
Bladder infection (Renal and urinary disorders) | 1
Ear infection (Ear and labyrinth disorders) | 1
Insomnia (General disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Night sweats (General disorders) | 1
Headache (Nervous system disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Soar throat (Gastrointestinal disorders) | 2
Boil in left axilla (Skin and subcutaneous tissue disorders) | 1
Left flank pain (General disorders) | 1
Seizure (Nervous system disorders) | 1
Skin rash (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Urinary urgency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT00503035/Prot_SAP_000.pdf